CLINICAL TRIAL: NCT07303868
Title: The Use of High Bile-Binding Foods to Reduce Upper Gastrointestinal Bile Acid Concentrations: A Novel Intervention for Children at Risk for Aspiration-Associated Complications (Aim 2)
Brief Title: The Use of High Bile-binding Foods to Reduce Upper Gastrointestinal Bile Acid Concentrations (Aim 2)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Rachel Rosen, Director, Aerodigestive Center, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00049734 Aim 2
Record Dates: First submitted 2025-03-29; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-03

CONDITIONS: Feeding Difficulties; Gastrostomy; Aspiration
Keywords: blenderized; bile acid; gastrostomy; aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low bile binding then high bile binding blenderized diets (Experimental): 2 weeks of low bile binding then 2 weeks of high bile binding blenderized diets
  Interventions: Drug: Low bile acid binding blenderized diet; Drug: High bile acid binding blenderized diet
- High bile binding then low bile binding blenderized diets (Experimental): 2 weeks of high bile binding then 2 weeks of low bile binding blenderized diets
  Interventions: Drug: Low bile acid binding blenderized diet; Drug: High bile acid binding blenderized diet
- amino acid-based formula (No Intervention): Observational arm

INTERVENTIONS:
Drug: Low bile acid binding blenderized diet — Low bile acid binding blenderized diet administered for 2 weeks
  Arms: High bile binding then low bile binding blenderized diets; Low bile binding then high bile binding blenderized diets
Drug: High bile acid binding blenderized diet — High bile acid binding blenderized diet administered for 2 weeks
  Arms: High bile binding then low bile binding blenderized diets; Low bile binding then high bile binding blenderized diets

SUMMARY:
Using a four-week randomized, crossover study design, we will assess the impact of 2 weeks of a high bile acid-binding blenderized diet, compared to 2 weeks of a low bile acid-binding blenderized diet, on gastric and salivary bile acid concentrations within individual participants. Four weeks of an amino acid formula will be a comparator group.

ELIGIBILITY:
Pediatric patients ages 5 to 21 in the randomized arm Inclusion criteria

* receive at least 80% of their nutritional needs via gastrostomy
* receive blenderized feeds or will start receiving blenderized feeds
* have no known allergies to ingredients in blenderized feeds;
* receive their bolus feeds within 30 minutes or less
* can receive their feeds by syringe push Exclusion criteria
* have undergone anti-reflux surgery
* receive post-pyloric feeds
* are allergic to any component of the administered diets
* cannot receive their gastrostomy feeds over 30 minutes
* require a feeding pump for feed administration (as the H-BBB is too thick for pump administration).

Pediatric patients ages 5 to 21 in the observational arm Inclusion

* receive at least 80% of their nutritional needs via gastrostomy
* are taking an amino acid formula
* have not undergone antireflux surgery Exclusion
* have undergone anti-reflux surgery
* receive post-pyloric feeds
* are not receiving an amino acid-based formula.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Gastric bile acid concentration | after 2 weeks on each of 2 diets (cross-over design)
  differences in total gastric bile acid concentrations at the end of each diet period

SECONDARY OUTCOMES:
Gastric bile acid concentration | after 2 weeks on each of 2 diets (cross-over design)
  changes in gastric bile acid composition (e.g., change in the proportion of gastric conjugated:unconjugated bile acid) between diet periods
Symptom scores | after 2 weeks on each of 2 diets (cross-over design)
  changes in symptoms over the two weeks between diet periods
Salivary and stool bile acid concentrations | after 2 weeks on each of 2 diets (cross-over design)
  changes in the total salivary and stool BA concentrations between diet periods;
Serum complement 4 (C4) | after 2 weeks on each of 2 diets (cross-over design)
  changes in serum C4 between diet periods
gastric, salivary, and stool bile acid | after 2 weeks on each of 2 diets (cross-over design)
  changes in gastric, salivary, and stool bile acid over time between the high bile binding blend, low bile binding blend and amino acid-based formula groups.

IPD SHARING:
Plan to Share IPD: No